CLINICAL TRIAL: NCT03296449
Title: Comparison Between Continuous Positive Airway Pressure and High-frequency Jet Ventilation in Nondependent Lung During One-lung Ventilation in Video-assisted Thoracoscopic Surgery
Brief Title: Comparison Between CPAP and HFJV During One-lung Ventilation in VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, María Galiana Ivars, Head of the Section of Clinical Anesthesia and Resuscitation, Hospital General Universitario de Alicante
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FREQUENCY
Record Dates: First submitted 2017-09-13; First posted 2017-09-28 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: One-Lung Ventilation; Thoracic Surgery, Video-Assisted
Keywords: Hypoxia; High-Frequency Jet Ventilation; Continuous Positive Airway Pressure
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- One-Lung Ventilation (No Intervention): During one-lung ventilation, when the chest is open, the non-dependent lung is collapsed and manipulated by the surgeon. It is the routine procedure during video-assisted thoracic surgery.
- CPAP to non-dependent lung (Active Comparator): The patient will be randomly assigned to the study arm "Continuous Positive Airway Pressure (CPAP)". CPAP will be applied for 20 minutes to the non-dependent lung at a pressure of 2-3cmH20 using the disposable Mallinckrodt Bronchocath CPAP system.
  Interventions: Procedure: CPAP
- HFJV to non-dependent lung (Experimental): The patient is randomly assigned to the study arm "High-frequency jet ventilation (HFJV)". HFJV will be applied for 20 minutes to the non-dependent lung with a driving pressure of a 0.6 atm, respiratory rate 100 cycles per minute using the Monsoone III Jet Ventilator (Acutronic, Hirzel, Switzerland).
  Interventions: Procedure: HFJV

INTERVENTIONS:
Procedure: CPAP — A recruitment maneuver will be applied to the ventilated lung. Immediately continuous positive airway pressure, at a pressure of 2-3cmH2O will applied to the non-ventilated lung for 20 minutes by the Mallinckrodt Bronchocath Disposable CPAP system (a recognised anesthetic breathing system design for CPAP).
  Arms: CPAP to non-dependent lung
Procedure: HFJV — A recruitment maneuver will be applied to the ventilated lung. Immediately, high-frequency jet ventilation, with a driving pressure of 0.5 atm and a respiratory rate of 100 cycles per minute will applied to the non-ventilated lung for 20 minutes using the Monsoone III Jet Ventilator (Acutronic, Hirzel, Switzerland). Monsoone III is a recognised ventilator design for HFJV.
  Arms: HFJV to non-dependent lung

SUMMARY:
This study compares two ventilatory techniques (continuous positive airway pressure vs high frequency jet ventilation) during one-lung ventilation (OLV) in video-assisted thoracic surgery (VATS). All patients were ventilated with both ventilatory techniques and parameters of gas exchange were determined through arterial blood gas test.

DETAILED DESCRIPTION:
One-lung ventilation is mandatory during most thoracic surgery procedures. During OLV, collapsed lung develops an intrapulmonary shunt leading to arterial hypoxemia. Since arterial hypoxemia is a critical intraoperative problem, many times , anesthesiologists have to use rescue ventilation strategies on non-dependent lung to improve arterial oxygen levels. The use of continuous positive airway pressure on non-dependent lung has become the most common technique to achieve that aim.

High-frequency jet ventilation on non-dependent lung may be considered as an alternative way of ventilation of the non-dependent lung during one-lung ventilation because it provides a suitable gaseous exchange while facilitating minimizing surgical field motion. However, this ventilation maneuver is rarely use by thoracic anesthesiologists.

Over the last years, video assisted thoracic surgery (VATS) has become widely utilized. This surgical technique becomes even more dependent on immobilization of the operation field than open-chest thoracic procedures. There is a lack of evidence in the current literature regarding the use of HFJV in VATS.

The purpose of this study is to evaluate the effects of HFJV as an alternative for the treatment of hypoxemia in VATS.

One-lung ventilation is mandatory during most thoracic surgery procedures. During OLV, collapsed lung develops an intrapulmonary shunt leading to arterial hypoxemia. Since arterial hypoxemia is a critical intraoperative problem, many times , anesthesiologists have to use rescue ventilation strategies on non-dependent lung to improve arterial oxygen levels. The use of continuous positive airway pressure on non-dependent lung has become the most common technique to achieve that aim.

High-frequency jet ventilation on non-dependent lung may be considered as an alternative way of ventilation of the non-dependent lung during one-lung ventilation because provide suitable gaseous exchange while facilitate minimizing surgical field motion. However , this ventilation maneuver is rarely use by thoracic anesthesiologists.

Over the last years, video assisted thoracic surgery (VATS) has become widely utilized. This surgical technique becomes even more dependent on immobilization of the operation field than open-chest thoracic procedures. There is a lack of evidence in the current literature about the use of HFJV in VATS.

The purpose of this study is to evaluate the effects of HFJV as an alternative for the treatment of hypoxemia in VATS.

ELIGIBILITY:
Inclusion Criteria:

* Subject requiring one-lung ventilation
* Subject under video-assisted thoracic surgery

Exclusion Criteria:

* Pregnant
* Emergent surgery
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 | 1 day
  Ratio of the arterial oxygen partial pressure (PaO2) to the inspired oxygen fraction (FiO2) determination.
  Time 0 (the patient is anesthetized and being ventilated on two lungs). Time 20 minutes (patient has been ventilated on one lung for 20 minutes). Time 40 minutes (following a period of 20 minutes on one intervention arm [either CPAP or HFJV]. The patient will then enter second intervention arm). Time 60 minutes ( 20 minutes after second intervention arm [either CPAP or HFJV])

SECONDARY OUTCOMES:
PaCO2 | 1 day
  Arterial carbon dioxide partial pressure determination. Time 0 (the patient is anesthetized and being ventilated on two lungs). Time 20 minutes (patient has been ventilated on one lung for 20 minutes). Time 40 minutes (following a period of 20 minutes on one intervention arm [either CPAP or HFJV]. The patient will then enter second intervention arm). Time 60 minutes ( 20 minutes after second intervention arm [either CPAP or HFJV])
Operative field conditions | 1 day
  Surgeon's subjective opinion about operating conditions during the interventions: impossible surgical access, acceptable operative filed or excellent operative field).
  Time 20 minutes (patient has been ventilated on one lung for 20 minutes). Time 40 minutes (following a period of 20 minutes on one intervention arm [either CPAP or HFJV]. The patient will then enter second intervention arm). Time 60 minutes ( 20 minutes after second intervention arm [either CPAP or HFJV])

OTHER OUTCOMES:
Airway pressures | 1 day
  Recording during mechanical ventilation of dependent lung airway pressures. Time 0 (the patient is anesthetized and being ventilated on two lungs). Time 20 minutes (patient has been ventilated on one lung for 20 minutes). Time 40 minutes (following a period of 20 minutes on one intervention arm [either CPAP or HFJV]. The patient will then enter second intervention arm). Time 60 minutes ( 20 minutes after second intervention arm [either CPAP or HFJV])
Adverse effects and complication | 30 days
  Any complication or adverse effect arising from ventilation techniques: need of intensive care unit admissions, re-intervention, or thoracotomy, surgical site infection, anastomosis leakage, and pneumonia.
Hemodynamic parameters | 1 day
  Heart rate and mean arterial blood pressure. Time 0 (the patient is anesthetized and being ventilated on two lungs). Time 20 minutes (patient has been ventilated on one lung for 20 minutes). Time 40 minutes (following a period of 20 minutes on one intervention arm [either CPAP or HFJV]. The patient will then enter second intervention arm). Time 60 minutes ( 20 minutes after second intervention arm [either CPAP or HFJV])

CONTACTS AND LOCATIONS:
Overall Officials: Maria Galiana, Principal Investigator — Hospital General Universitario de Alicante
Locations (1):
- Hospital General Universitario de Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided